CLINICAL TRIAL: NCT00451113
Title: Sitagliptin in the Elderly
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Merck Frosst Canada Ltd. (Industry)
Responsible Party: Principal Investigator, Graydon Meneilly, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: H06-03067
Record Dates: First submitted 2007-03-21; First posted 2007-03-23 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes; Older adults; Incretins; Hyperglycemia; Insulin resistance
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperglycemia; Insulin Resistance | interventions — Sitagliptin Phosphate; Dipeptidyl-Peptidase IV Inhibitors

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Sitagliptin 100 mg — All subjects will receive a single 100 mg dose of sitagliptin and a placebo. Which they are given first is determined randomly.
  Other Names: Januvia; MK-0431; Dipeptidyl peptidase IV inhibitor (DPP-4 inhibitor)

SUMMARY:
Diabetes is common in the elderly; by the age of 70, approximately 25% of the population will have diabetes. Unfortunately, currently available medications are often not as effective or not well tolerated in older adults. Sitagliptin is a new medication in a new class of agent called incretins. Incretins have many potential advantages for the treatment of diabetes in the elderly. They stimulate insulin secretion, which is impaired in all older people with diabetes. The incidence of hypoglycemia with currently available medications increases with age, and incretins rarely cause hypoglycemia . They assist with weight loss, whereas many current medications used to manage diabetes result in weight gain in the elderly. They improve insulin action, and insulin resistance is a major problem in older people with diabetes.

DETAILED DESCRIPTION:
To date, no clinical trials have been conducted specifically in the elderly, but the data noted above from our laboratory would imply that inhibitors of this enzyme could be more effective in the elderly patient population. In addition, we have convincingly demonstrated that diabetes in the elderly is metabolically distinct from diabetes in middle aged patients (1). Thus, it is clear further studies are warranted to determine the effectiveness of drugs in this class in elderly patients with diabetes. We propose a series of studies with your DP4 inhibitor sitaglipitin to determine its efficacy and safety in an elderly patient population with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes managed by diet or metformin only
* A1c < 8.5%

Exclusion Criteria:

* treated with insulin or oral agents other than metformin in the past 6 months
* evidence of diabetic complications including coronary artery disease, stroke, transient ischemic attacks, peripheral vascular disease, nephropathy, retinopathy, or neuropathy
* type 1 diabetes or a history suggestive of a secondary causes of diabetes
* A1c ≥ 8.5%
* participated in another clinical trial within the past 30 days

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 12 (Actual)
Dates: Start 2006-11; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Safety and efficacy of Sitagliptin in an elderly population with type 2 diabetes

CONTACTS AND LOCATIONS:
Overall Officials: Graydon Meneilly, MD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia Gerontology & Diabetes Research Centre, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Stafford S, Elahi D, Meneilly GS. Effect of the dipeptidyl peptidase-4 inhibitor sitagliptin in older adults with type 2 diabetes mellitus. J Am Geriatr Soc. 2011 Jun;59(6):1148-9. doi: 10.1111/j.1532-5415.2011.03438.x. No abstract available. PMID 21668924